CLINICAL TRIAL: NCT01375998
Title: Drug Use Investigation of YAZ
Brief Title: YAZ Post-marketing Surveillance in Japan
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 15328; YAZ-DUI (Other: Company internal)
Record Dates: First submitted 2011-06-08; First posted 2011-06-20 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Dysmenorrhea
Keywords: YAZ; Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: EE20/DRSP(YAZ, BAY86-5300)

INTERVENTIONS:
Drug: EE20/DRSP(YAZ, BAY86-5300) — Patients in daily life treatment receiving YAZ for dysmenorrhea.

SUMMARY:
This study is a regulatory post marketing surveillance in Japan, and it is a local prospective and observational study of patients who have received YAZ for dysmenorrhea. The objective of this study is to assess safety and efficacy of using YAZ in clinical practice. A total 3,000 patients will be recruited and followed 3 years since starting YAZ administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received YAZ for dysmenorrhea Additional criteria for QOL questionnaire
* Patient informed consent

Exclusion Criteria:

* Patients who are contraindicated based on the product label Additional criteria for QOL questionnaire
* Six months or less after treatment of estrogen or estrogen combination drug

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target population of this study is patients who have received a prescription of YAZ on the basis of the decision of the treating gynecologist. The study is expected to collect data of 3,000 patients in about 300 gynecological practices in Japan.
Sampling Method: Non-Probability Sample
Enrollment: 3273 (Actual)
Dates: Start 2011-06-09 (Actual); Primary Completion 2017-12-05 (Actual); Study Completion 2018-03-08 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions and sever adverse events | During YAZ administration, up to 3 years
Change from baseline in severity of dysmenorrhea at 6th cycles (28 days per cycle) | Baseline and during YAZ administration, up to 3 years

SECONDARY OUTCOMES:
Incidence of adverse events | During YAZ administration, up to 3 years
Unpleasant physical symptoms collection | Baseline and during YAZ administration, up to 3 years
Unpleasant psychological symptoms collection | Baseline and during YAZ administration, up to 3 years
Analgesic drug for dysmenorrhea | During YAZ administration, up to 3 years
QOL survey using Short-Form 36-Item Health Survey (SF-36) | Baseline and at 6th - 8th cycles (28 datys per cycle)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Japan

REFERENCES:
- [Derived] Momoeda M, Akiyama S, Tanaka K, Suzukamo Y. Quality of Life in Japanese Patients with Dysmenorrhea Treated with Ethinylestradiol 20 mug/Drospirenone 3 mg in a Real-World Setting: An Observational Study. Int J Womens Health. 2020 May 4;12:327-338. doi: 10.2147/IJWH.S238460. eCollection 2020. PMID 32440228